CLINICAL TRIAL: NCT07132645
Title: An Exploratory Study of [68Ga]Ga-Fibroblast Activation Protein Inhibitor 4 ([68Ga]Ga-FAPI-04) in Patients With High-Grade Neuroendocrine Neoplasms
Brief Title: An Investigational Scan ([68Ga] Ga-FAPI-04 PET/CT) for the Imaging of Patients With High-Grade Neuroendocrine Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Neuroendocrine Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UMCC 2024.069; NCI-2025-04557 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00237403 (Other: University of Michigan)
Record Dates: First submitted 2025-07-14; First posted 2025-08-20 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 68Ga-FAPI; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Basic science ([68Ga] Ga-FAPI-04) (Experimental): Patients receive [68Ga] Ga-FAPI-04 IV, followed 1 hour later by PET/CT scan over approximately 25 minutes.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68-DOTA-FAPI-04; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Gallium Ga 68-DOTA-FAPI-04 — Given IV
  Other Names: 68Ga-DOTA-FAPI-04; 68Ga-FAPi-04; GALLIUM GA-68-DOTA-FAPI-04; Gallium-68-FAPi-04
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This early phase I trial determines where and to what degree the tracer [68Ga] Ga-FAPI-04 accumulates in normal and cancer tissues in patients with high grade neuroendocrine cancer. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research [68Ga] Ga-FAPI-04. Because some cancers take up [68Ga] Ga-FAPI-04, it can be seen with PET. CT utilizes x-rays that traverse body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in patient's body.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Current neuroendocrine tumor diagnosis AND high-grade neuroendocrine tumor presentation determined using the following criteria(s):

  * Previous low uptake of [68Ga] Ga-DOTATATE PET/CT scan OR
  * Krenning Score ≥ 3 OR
  * Ki67 index ≥ 20%
* Able to lie flat for 60 minutes
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Patient recently underwent surgery with wound healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of Gallium Ga 68-DOTA-FAPI-04 ([68Ga]Ga-FAPI-04) | Day 1
Pharmacokinetics of [68Ga] Ga-FAPI-04 | Day 1
  We will monitor/measure the amount of Ga-FAPI-04 seen within different tissue in patients that have neuroendocrine tumors. We will specifically measure the ratio of uptake in the tumors in comparison to reference tissues such as liver or muscle.

SECONDARY OUTCOMES:
Tissue concentrations of [68Ga] Ga-FAPI-04 retention in tumors | Day 1
Standardized uptake values (SUV) of [68Ga] Ga-FAPI-04 retention in tumors | Day 1
  Will compare the difference in SUVmax uptake within each subject using a two-side, one-sample t-test.
Clinical diagnostic performance of [68Ga] Ga-FAPI-04 | Day 1
  When a comparison Ga-DOTATATE scan is available, we will look at the uptake in the tumor in the SOC image related to reference tissue and then compare the FAPI-04 uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Viglianti, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided